CLINICAL TRIAL: NCT03042455
Title: Combined Repetitive Transcranial Magnetic Stimulation and Robot-Assisted Upper Arm Training in Subacute Stroke Patients : Randomized Controlled Trial
Brief Title: Combined Repetitive Transcranial Magnetic Stimulation and Robot-Assisted Upper Arm Training in Subacute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1-2014-0083
Record Dates: First submitted 2017-01-30; First posted 2017-02-03 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Robot and rTMS (Experimental): Robot-Assisted upper arm training and Repetitive Transcranial Magnetic Stimulation group(intervention group 1)
  Interventions: Device: Armeo and rTMS
- Robot (Experimental): Robot-Assisted upper arm training group(intervention group2)
  Interventions: Device: Armeo
- Conventional (Active Comparator): Conventional training group(control group)
  Interventions: Other: Control group

INTERVENTIONS:
Device: Armeo and rTMS — The Armeo, a robot with a spring mechanism allowing adjustable arm weight support, can generate assistive forces of up to 66N in flexion/extension and up to 30N for the arm and forearm respectively. This robot integrates seven angle sensors and one pressure sensor that allow direct interaction between the motion of the patient's arm and the associated therapy software. rTMS is a magnetic method used to stimulate small regions of the brain.
  The Robot and rTMS group will receive the robot-assisted upper arm training and rTMS for 5 times per week, for 4 weeks. And all patients of three groups will receive the additional conventional occupational therapy for 30 minutes daily 5 times per week, for 4 weeks.
  Other Names: Robot-Assisted upper arm training(Armeo); Repetitive Transcranial Magnetic Stimulation(rTMS)
  Arms: Robot and rTMS
Device: Armeo — The Armeo, a robot with a spring mechanism allowing adjustable arm weight support, can generate assistive forces of up to 66N in flexion/extension and up to 30N for the arm and forearm respectively. This robot integrates seven angle sensors and one pressure sensor that allow direct interaction between the motion of the patient's arm and the associated therapy software. The Robot group will receive the robot-assisted upper arm training for 30 minutes daily 5 times per week, for 4 weeks. And all patients of three groups will receive the additional conventional occupational therapy for 30 minutes daily 5 times per week, for 4 weeks.
  Other Names: Robot-Assisted upper arm training(Armeo)
  Arms: Robot
Other: Control group — The conventional group will receive occupational therapy for 30 minutes daily 5 times per week, for 4 weeks instead of Robot or rTMS. And all patients of three groups will receive the additional conventional occupational therapy for 30 minutes daily 5 times per week, for 4 weeks.
  Other Names: conventional training
  Arms: Conventional

SUMMARY:
This study was designed to establish the clinical evidence for effect of Robot-Assisted upper arm training and Repetitive Transcranial Magnetic Stimulation on upper limb function of subacute stroke patients.

* Purpose : to elucidate the effect of Robot-Assisted upper arm training and Repetitive Transcranial Magnetic Stimulation on upper limb function of stroke patients compared to conventional occupational therapy
* Subjects : total 99 patients with stroke whose upper limb functions are impaired
* Intervention : 4 weeks of therapy (5 days per week)
* Studies : upper limb functional assessment (FMA, MFT, WMFT), computerized motion analysis
* Evaluation plan : 1) pre-intervention, 2) post-2 weeks of intervention, 3) post-4 weeks of intervention, 4) 4 weeks after end of intervention

ELIGIBILITY:
Inclusion Criteria:

* Upper FMA 7-38
* Hemiplegic patients within 6months after stroke onset
* male or female, 20 years older

Exclusion Criteria:

* Patients with cognitive impairment who are unable to comply with protocol-required procedure
* Quadriplegic or double hemiplegic patients
* Patients with musculoskeletal disease, peripheral nerve disease in upper extremity
* Patients with lower motor neuron disease
* Patients who cannot perform rTMS
* Pregnant woman

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-06-18 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | 1 minute before the first intervention
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia.
Fugl-Meyer Assessment (FMA) | 2 weeks after the first intervention
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia.
Fugl-Meyer Assessment (FMA) | 4 weeks after the first intervention
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia.
Fugl-Meyer Assessment (FMA) | 4 weeks after the final intervention
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia.

SECONDARY OUTCOMES:
Wolf motor function test | 1 minute before the first intervention
  The Wolf Motor Function Test (WMFT) is a quantitative index of upper extremity motor ability examinable through the use of timed and functional tasks.
Wolf motor function test | 2 weeks after the first intervention
  The Wolf Motor Function Test (WMFT) is a quantitative index of upper extremity motor ability examinable through the use of timed and functional tasks.
Wolf motor function test | 4 weeks after the first intervention
  The Wolf Motor Function Test (WMFT) is a quantitative index of upper extremity motor ability examinable through the use of timed and functional tasks.
Wolf motor function test | 4 weeks after the final intervention
  The Wolf Motor Function Test (WMFT) is a quantitative index of upper extremity motor ability examinable through the use of timed and functional tasks.
Manual Function test | 1 minute before the first intervention
  The Manual Function Test (MFT) was developed to evaluate unilateral manual performance in hemiparetic patients after stroke.
Manual Function test | 2 weeks after the first intervention
  The Manual Function Test (MFT) was developed to evaluate unilateral manual performance in hemiparetic patients after stroke.
Manual Function test | 4 weeks after the first intervention
  The Manual Function Test (MFT) was developed to evaluate unilateral manual performance in hemiparetic patients after stroke.
Manual Function test | 4 weeks after the final intervention
  The Manual Function Test (MFT) was developed to evaluate unilateral manual performance in hemiparetic patients after stroke.
Kinematic data of computerized 3D motion analysis | 1 minute before the first intervention
  D motion analysis will be performed using a computerized motion analysis system (VICON MX-T10 System with 6 infrared cameras, Oxford Metrics Inc., Oxford, UK) to measure the kinematic data (angle of each joint) during the task of drinking from a cup
Kinematic data of computerized 3D motion analysis | 2 weeks after the first intervention
  D motion analysis will be performed using a computerized motion analysis system (VICON MX-T10 System with 6 infrared cameras, Oxford Metrics Inc., Oxford, UK) to measure the kinematic data (angle of each joint) during the task of drinking from a cup
Kinematic data of computerized 3D motion analysis | 4 weeks after the first intervention
  D motion analysis will be performed using a computerized motion analysis system (VICON MX-T10 System with 6 infrared cameras, Oxford Metrics Inc., Oxford, UK) to measure the kinematic data (angle of each joint) during the task of drinking from a cup
Kinematic data of computerized 3D motion analysis | 4 weeks after the final intervention
  D motion analysis will be performed using a computerized motion analysis system (VICON MX-T10 System with 6 infrared cameras, Oxford Metrics Inc., Oxford, UK) to measure the kinematic data (angle of each joint) during the task of drinking from a cup

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Medicine, Severance Hospital, Research Institute of Rehabilitation Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided